CLINICAL TRIAL: NCT05373706
Title: Development and Preliminary Examination of Two Brief Personalized Feedback Interventions Focused on Lab-based and EMA Alcohol Cues to Reduce Hazardous Young Adult Alcohol Use
Brief Title: Testing Brief Personalized Feedback Integrating EMA Alcohol Cue Information
Acronym: Project ACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Jason Ramirez, Research Assistant Professor: School of Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00014778; 1R34AA027302-01A1 (NIH)
Record Dates: First submitted 2022-05-09; First posted 2022-05-13 (Actual); Results first posted 2024-06-04 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Alcohol Drinking; Problem Drinking
Keywords: Alcohol; Intervention; Young Adults; Personalized Feedback
MeSH Terms: conditions — Alcohol Drinking; Alcoholism | interventions — Ethanol

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two conditions (Personalized feedback and assessment-only control group).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cue Reactivity Personalized Feedback Intervention (PFI) (Experimental): Participants randomized to the Cue Reactivity PFI condition will receive personalized feedback at the end of completing 17 days of ecological momentary assessments (EMAs) four times a day. The personalized feedback will be delivered online and contains information summarizing participants' desire to drink as it varied as a function of several real-world factors across the 17-day EMA period.
  Interventions: Behavioral: Alcohol Cue Reactivity Personalized Feedback Intervention
- Assessment-only control (No Intervention): Participants randomized to the control group will not receive any intervention. They will be an assessment-only control group.

INTERVENTIONS:
Behavioral: Alcohol Cue Reactivity Personalized Feedback Intervention — This online brief intervention provides personalized feedback using EMA data focused on alcohol cue reactivity to reduce alcohol misuse among young adults.
  Arms: Cue Reactivity Personalized Feedback Intervention (PFI)

SUMMARY:
This study aims to develop a brief intervention that incorporates ecological momentary assessments (EMAs; i.e., four brief surveys per day for 17 days) to create personalized feedback targeting high-risk alcohol use among young adult drinkers. The intervention mainly focuses on providing feedback on individuals' drinking desire and how it varies as a function of a number of real-world factors. Other psycho-educational alcohol-related content is also provided in the intervention including strategies for decreasing exposure to cues that increase drinking desires and how to cope with increased desire to drink. This brief intervention will be used in a randomized controlled trial (RCT) comparing young adults who receive the intervention with those who only complete identical assessments.

DETAILED DESCRIPTION:
The purpose of this study is to develop and test a brief intervention that provides personalized feedback to young adults using participants' own event-level, real-world experiences. The aim of the intervention is to increase young adults' awareness of their desire to drink as it varies as a function of a number of real-world factors including alcohol cues, social context, physical context, anticipation of later drinking, mood, and time of day. The intervention also aims to equip young adults with strategies for reducing exposure to factors that increase their desire to drink, how to cope with an increased desire to drink, and how to reduce potential harms from drinking.

This brief personalized feedback intervention is used in a randomized controlled trial comparing young adults who receive the intervention with those who complete the EMAs but do not receive any personalized feedback. Assessments include an eligibility survey, baseline assessment, 17 days of EMAs (4x/day), and follow-up assessments occurring 2-weeks and 3-months post-intervention. The 2-week and 3-month follow-ups occurred 2-weeks and 3-months, respectively, from Day 17 of the EMA period, because the intervention was delivered on Day 17. The intervention will be examined for its feasibility, acceptability, and its effects in reducing alcohol-related outcomes at the follow-up assessments.

ELIGIBILITY:
Inclusion Criteria:

* 1) Between ages 18-24, 2) Lives in Washington state, 3) Reports drinking at least two days per week in the last six months, 4) Reports at least one heavy drinking episode (4+/5+ drinks for women/men) in the past month, 5) Open to changing drinking behavior, 6) Schedule allows for participation in study with daily surveys, 7) Able to attend Zoom training session, 8) Must have cellphone for daily surveys.

Exclusion Criteria:

* 1) Actively seeking treatment for alcohol use, 2) Currently participating in another study in our research center regarding young adult drinking behavior.

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 99 (Actual)
Dates: Start 2022-04-29 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Ramirez, PhD, Principal Investigator — University of Washington; Anne Fairlie, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
We plan to share limited, de-identified datasets for the purposes of data analysis and dissemination.
Supporting Information: SAP, Analytic Code
Time Frame: Data dictionaries and limited datasets can be made available starting in February 2023.
Access Criteria: Individual requests to access data with intended purpose should be made to Drs. Fairlie and Ramirez and will be reviewed by the investigative team.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from Washington state using a variety of recruitment methods (e.g., predominantly Instagram, random selection of students from university registrar's lists). Individuals were invited to complete an online eligibility survey for participation in a randomized clinical trial to test the effect of an online personalized feedback intervention. Recruitment/enrollment period went from April 2022 to January 2023.
Period: Overall Study
Arm/Group | Assessment-only Control | Cue Reactivity Personalized Feedback Intervention (PFI)
Started | 48 | 51
Completed | 46 | 49
Not Completed | 2 | 2
Not completed — Lost to Follow-up | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Assessment-only Control | Cue Reactivity Personalized Feedback Intervention (PFI) | Total
Number analyzed (Participants) | 48 | 51 | 99
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 48 | 51 | 99
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.42 (1.75) | 21.69 (1.86) | 21.56 (1.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 28 | 54
  Male | 22 | 23 | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 5 | 7
  Not Hispanic or Latino | 46 | 46 | 92
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 7 | 10 | 17
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 3 | 1 | 4
  White | 30 | 34 | 64
  More than one race | 6 | 3 | 9
  Unknown or Not Reported | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 48 | 51 | 99
Current educational status [Count of Participants; unit: Participants] — Currently a 4-year college/university student versus not
  Participants
    4-year student | 27 | 28 | 55
    Not a 4-year student | 21 | 23 | 44

OUTCOME MEASURES:

1. Primary Outcome: Daily Drinking Questionnaire
Description: Number of standard drinks consumed on each day of a typical week during the [past 3 months for baseline and 3-month follow-up; past two weeks for 2-week follow-up]. Participants responded on a scale from 0 (0 drinks) to 25 (25 or more drinks). Totals for each day are summed to calculate the typical number of drinks consumed per week.
Time Frame: Baseline, 2 week follow-up, and 3 month follow-up
Population: Young adults
Measure: Mean (Standard Deviation); unit: Drinks per week
Arm/Group | Assessment-only Control | Cue Reactivity Personalized Feedback Intervention (PFI)
Number analyzed (Participants) | 48 | 51
Drinks per week
  Baseline | 12.23 (11.85) | 11.78 (7.24)
  2-Week Follow-Up | 10.31 (10.77) | 9.40 (6.28)
  3-Month Follow-Up | 7.54 (7.16) | 8.49 (7.16)
Statistical Analysis 1: Comparison: Assessment-only Control vs Cue Reactivity Personalized Feedback Intervention (PFI); Changes from Baseline to 2-Week Follow-Up for PFI versus AOC reported in this section; Test type: Superiority — Generalized linear mixed model was estimated using a sample of N=99 with a Condition × 2-Week Follow-Up interaction. AOC was the reference category for Condition, and Baseline was the reference category for 2-Week Follow-Up; p = 0.68, Generalized linear mixed model; Models controlled for sex assigned at birth, age, and student status (4-year vs. not) and used a Poisson error distribution; Count/Rate Ratio = 0.95, 95% CI 2-sided [0.76 to 1.20]
Statistical Analysis 2: Comparison: Assessment-only Control vs Cue Reactivity Personalized Feedback Intervention (PFI); Changes from Baseline to 3-Month Follow-Up for PFI versus AOC reported in this section; Test type: Superiority — Generalized linear mixed model was estimated using a sample of N=99 with a Condition × 3-Month Follow-Up interaction. AOC was the reference category for Condition, and Baseline was the reference category for 3-Month Follow-Up; p = 0.56, Generalized linear mixed model; [statistical method as in outcome 1, analysis 1]; Count/Rate Ratio = 1.10, 95% CI 2-sided [0.81 to 1.49]

2. Primary Outcome: Number of Heavy Episodic Drinking Occasions
Description: Participants were asked, "During the past two weeks, how many times did you have [4/5 for females/males] or more drinks at one sitting?". Participants responded on a scale from 0 (0 times) to 10 (10 or more times) and possible range was 0-10.
Time Frame: Baseline, 2 week follow-up, and 3 month follow-up
Population: Young adults
Measure: Mean (Standard Deviation); unit: Number heavy episodic drinking occasions
Arm/Group | Assessment-only Control | Cue Reactivity Personalized Feedback Intervention (PFI)
Number analyzed (Participants) | 48 | 51
Number heavy episodic drinking occasions
  Baseline | 2.46 (2.32) | 2.43 (1.97)
  2-Week Follow-Up | 2.46 (2.10) | 2.28 (1.72)
  3-Month Follow-Up | 1.63 (1.82) | 1.98 (1.93)
Statistical Analysis 1: Comparison: Assessment-only Control vs Cue Reactivity Personalized Feedback Intervention (PFI); Changes from Baseline to 2-Week Follow-Up for PFI versus AOC reported in this section; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.68, Generalized linear mixed model; [statistical method as in outcome 1, analysis 1]; Count/Rate Ratio = 0.93, 95% CI 2-sided [0.64 to 1.33]
Statistical Analysis 2: Comparison: Assessment-only Control vs Cue Reactivity Personalized Feedback Intervention (PFI); Changes from Baseline to 3-Month Follow-Up for PFI versus AOC reported in this section; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p = 0.30, Generalized linear mixed model; [statistical method as in outcome 1, analysis 1]; Count/Rate Ratio = 1.24, 95% CI 2-sided [0.82 to 1.88]

3. Primary Outcome: Penn Alcohol Craving Scale
Description: Self-reported subjective alcohol craving during the past week. Response options were scored from "0" to "6" with text varying across items. A sum score of the five items was calculated and the possible range was from 0-30. Higher scores reflect more craving.
Time Frame: Baseline, 2 week follow-up, and 3 month follow-up
Population: Young adults
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Assessment-only Control | Cue Reactivity Personalized Feedback Intervention (PFI)
Number analyzed (Participants) | 48 | 51
Score on a scale
  Baseline | 6.58 (5.12) | 7.92 (5.07)
  2-Week Follow-Up | 7.80 (4.55) | 8.66 (5.81)
  3-Month Follow-Up | 5.80 (4.28) | 7.46 (5.01)
Statistical Analysis 1: Comparison: Assessment-only Control vs Cue Reactivity Personalized Feedback Intervention (PFI); Changes from Baseline to 2-Week Follow-Up for PFI versus AOC reported in this section; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.36, Generalized linear mixed model; [statistical method as in outcome 1, analysis 1]; Count/Rate Ratio = 0.89, 95% CI 2-sided [0.69 to 1.15]
Statistical Analysis 2: Comparison: Assessment-only Control vs Cue Reactivity Personalized Feedback Intervention (PFI); Changes from Baseline to 3-Month Follow-Up for PFI versus AOC reported in this section; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p = 0.73, Generalized linear mixed model; [statistical method as in outcome 1, analysis 1]; Count/Rate Ratio = 1.05, 95% CI 2-sided [0.80 to 1.38]

4. Primary Outcome: Brief Young Adult Alcohol Consequences Questionnaire
Description: Participants responded "no" (0) or "yes" (1) to whether they experienced each of 24 consequences during the [past 3 months for baseline and 3-month follow-up; past two weeks for 2-week follow-up]. A sum of the number of negative alcohol-related consequences was calculated and the possible range was 0-24.
Time Frame: Baseline, 2 week follow-up, and 3 month follow-up
Population: Young adults
Measure: Mean (Standard Deviation); unit: Number of consequences (range 0-24)
Arm/Group | Assessment-only Control | Cue Reactivity Personalized Feedback Intervention (PFI)
Number analyzed (Participants) | 48 | 51
Number of consequences (range 0-24)
  Baseline | 7.81 (5.02) | 8.78 (4.13)
  2-Week Follow-Up | 4.78 (4.35) | 4.52 (3.61)
  3-Month Follow-Up | 6.37 (5.65) | 6.04 (5.12)
Statistical Analysis 1: Comparison: Assessment-only Control vs Cue Reactivity Personalized Feedback Intervention (PFI); Changes from Baseline to 2-Week Follow-Up for PFI versus AOC reported in this section; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.11, Generalized linear mixed model; [statistical method as in outcome 1, analysis 1]; Count/Rate Ratio = 0.83, 95% CI 2-sided [0.66 to 1.04]
Statistical Analysis 2: Comparison: Assessment-only Control vs Cue Reactivity Personalized Feedback Intervention (PFI); Changes from Baseline to 3-Month Follow-Up for PFI versus AOC reported in this section; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p = 0.38, Generalized linear mixed model; [statistical method as in outcome 1, analysis 1]; Count/Rate Ratio = 0.88, 95% CI 2-sided [0.66 to 1.17]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected between initial screening and final follow-up for each participant, a period of approximately 4 months.
Description: We used clinicaltrials.gov definitions for adverse events and serious adverse events.
Arm/Group | Assessment-only Control | Cue Reactivity Personalized Feedback Intervention (PFI)
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/51
Other Adverse Events (participants affected / at risk) | 0/48 | 0/51

LIMITATIONS AND CAVEATS:
This is a small pilot trial designed to collect feasibility and acceptability information. Study data were collected during the COVID-19 pandemic from April 2022 through May 2023, which may have impacted alcohol use and contexts of alcohol use among young adult participants. All findings are based on self-report of alcohol use.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2024-04-30): https://cdn.clinicaltrials.gov/large-docs/06/NCT05373706/Prot_000.pdf
  • Statistical Analysis Plan (2024-04-30): https://cdn.clinicaltrials.gov/large-docs/06/NCT05373706/SAP_001.pdf
  • Informed Consent Form (2022-02-03): https://cdn.clinicaltrials.gov/large-docs/06/NCT05373706/ICF_002.pdf